CLINICAL TRIAL: NCT02512003
Title: Pilot Study of the REVA Sirolimus-Eluting Bioresorbable Coronary Scaffold
Brief Title: Pilot Study of the Fantom Bioresorbable Scaffold (FANTOM I)
Acronym: FANTOM I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: REVA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCT6000
Record Dates: First submitted 2015-07-14; First posted 2015-07-30 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fantom Treatment group (Experimental)
  Interventions: Device: Fantom Scaffold

INTERVENTIONS:
Device: Fantom Scaffold

SUMMARY:
The FANTOM I pilot study is intended to assess safety of the Fantom Bioresorbable Coronary Scaffold in native coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

* Patient has evidence of myocardial ischemia or a positive functional study
* Patient has a normal CK-MB
* Target lesion has a visually estimated stenosis of ≥50% and <100%
* Target lesion is located in a native coronary artery with average reference vessel diameter ≥ 2.7mm and ≤ 3.3mm
* Target lesion length must be ≤ 14mm

Exclusion Criteria:

* Patient has experienced a myocardial infarction (CK-MB or Troponin > 5 X ULN) within 72 hours of the procedure
* Patient has a left ventricular ejection fraction < 25%
* Patient has unprotected lest main coronary disease with ≥50% stenosis
* The target vessel is totally occluded (TIMI Flow 0 or 1)
* Target lesion involves a bifurcation (a lesion with a side branch ≥ 2.0 mm in diameter containing a ≥ 50% stenosis).
* Target lesion is located within a bypass graft
* Target lesion has possible or definite thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Ischemia-driven Target Lesion Revascularization (TLR) | 4 months
  Percent of Patients with TLR at 4 months

SECONDARY OUTCOMES:
Quantitative Coronary Angiography (QCA) derived parameters | 4 months
  Late Loss
Quantitative Coronary Angiography (QCA) derived parameters | 4 months
  Restenosis Rate
Quantitative Coronary Angiography (QCA) derived parameters | 4 months
  % Diameter Stenosis
Quantitative Coronary Angiography (QCA) derived parameters | 4 months
  Minimum Lumen Diameter
Quantitative Coronary Angiography (QCA) derived parameters | 4 months
  Neointimal Volume
Intravascular Ultrasound (IVUS) derived parameters | 4 months
  Late Loss
Intravascular Ultrasound (IVUS) derived parameters | 4 months
  Restenosis Rate
Intravascular Ultrasound (IVUS) derived parameters | 4 months
  % Diameter Stenosis
Intravascular Ultrasound (IVUS) derived parameters | 4 months
  Minimum Lumen Diameter
Intravascular Ultrasound (IVUS) derived parameters | 4 months
  Neointimal Volume
Major Adverse Cardiac Events | 12, 24, 36, 48 and 60 months
  Death, Q-Wave Myocardial Infarction, Non Q-Wave Myocardial Infarction (CK-MB > 5x normal), Target Vessel Revascularization
Target Lesion Revascularization (TLR) | 12, 24, 36, 48 and 60 months
  Percentage of patients with TLR at each time point
Target Vessel Revascularization | 12, 24, 36, 48 and 60 months
  Percentage of patients with TVR at each time point
Target Vessel Failure (TVF) | 12, 24, 36, 48 and 60 months
  Percentage of patients with TVF at each time point
Acute Technical Success | Day 0
  Percentage of patients with successful acute delivery and deployment of the device
Procedural Success | 30 days
  Percentage of patients with angiographic success (final diameter stenosis <50% without occurrence of MACE)
Optical Coherence Tomography (OCT) Imaging on a Subset of Patients | 4 months
  Qualitative measures in a subset of patients

CONTACTS AND LOCATIONS:
Locations (2):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, Brazil
- Pracownia Kardiologii Inwazyjnej I Katedry i Kliniki Kardiologii WUM, Warsaw, Poland